CLINICAL TRIAL: NCT03280199
Title: The Impact of Different Simulator Characteristics on Transfer of Learning
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Was not feasible
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Martin G. Tolsgaard, MD PhD, assistant professor., Rigshospitalet, Denmark
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 2017-09-GCMT
Record Dates: First submitted 2017-09-10; First posted 2017-09-12 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Simulation-based Medical Education; Ultrasound Simulation; Education, Professional

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Type of simulator - 1 (Other): VR simulator with physical mannequin and probe.
  PLEASE NOTE THAT THE INTERVENTIONS BEING COMPARED ARE DIFFERENT TYPES OF SIMULATORS - NOT A DRUG!
  Interventions: Other: simulation types
- Type of simulator - 2 (Other): VR simulator with virtual mannequin / abdomen
  PLEASE NOTE THAT THE INTERVENTIONS BEING COMPARED ARE DIFFERENT TYPES OF SIMULATORS - NOT A DRUG!
  Interventions: Other: simulation types
- Type of image acquisition - 3 (Other): US images are acquired through real US volumes from patients
  PLEASE NOTE THAT THE INTERVENTIONS BEING COMPARED ARE DIFFERENT TYPES OF SIMULATORS - NOT A DRUG!
  Interventions: Other: simulation types
- Type of image acquisition - 4 (Other): US images are acquired through computer-generated images.
  PLEASE NOTE THAT THE INTERVENTIONS BEING COMPARED ARE DIFFERENT TYPES OF SIMULATORS - NOT A DRUG!
  Interventions: Other: simulation types

INTERVENTIONS:
Other: simulation types — Different types of simulation interfaces and image acquisitions

SUMMARY:
This study aims to explore the impact of different simulator characteristics on transfer of learning.

DETAILED DESCRIPTION:
During an ISUOG basic training course, participants will be randomly assigned to 30 minutes of simulator training during which time they will practice the 2nd trimester US scan. A total of four different simulators are being used for training. After completing the practical basic training session, they shift the type of simulator that they trained on to one of the remaining three simulators. On this simulator, they are required to perform selected planes for the 2nd-trimester scan. The planes produced are recorded and evaluated by fetal medicine specialists using the ISUOG 20 planes checklist. The performances of participants coming from each of the four simulators are examined and the role of 1) type of simulator interaction (physical mannequin vs. virtual abdomen vs. fixed-point scan) and 2) the type of image acquisition (real US images vs. computer-generated images) are examined.

ELIGIBILITY:
Inclusion Criteria:

ISUOG course participants

Exclusion Criteria:

More than 50 independent 2nd trimester US scan before attending the course.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Correct planes | 30 minutes
  Number of correct planes produced

IPD SHARING:
Plan to Share IPD: No